CLINICAL TRIAL: NCT06522490
Title: Effects of Virtual Discrete Trial Training on Children With Autism Spectrum Disorder
Acronym: VDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU-123 Shahzadi Arshad
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Video Training was used for the experimental group
  Interventions: Other: Virtual discrete trial training
- Controlled group (Active Comparator): Face to face therapy was used for the control group
  Interventions: Other: Virtual discrete trial training

INTERVENTIONS:
Other: Virtual discrete trial training — VDT was given to Experimental group.
  Other Names: Face to face therapy

SUMMARY:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder categorized by deficits in social communication and the occurrence of restricted interests and repetitive behaviors. The cautionary needs of children with ASD are significant, it affects parents and siblings as well and requires substantial social support. If adequate intervention is not provided to children with ASD on time, then they may face many difficulties for example in academic work. They face social isolation and may develop additional challenging behaviors. Applied behavior analysis (ABA) is one of the most commonly used supported treatments for autism spectrum disorder. Discrete Trial Training (DTT) is one of the most structured Applied Behavior Analysis (ABA) types. DTT is the best standardized therapy for ASD. The ABA explores human interactions with their environment over time and develops interventional strategies to diminish the decline in the troublesomeness of social behavior among individuals with ASD. DTT through video training Program will be an effective in improving the communication skills of children with ASD. The video training program offers excellent accessibility and is inexpensive because it can be administered remotely and at home as well. It also reduces the resource barrios.

A randomized controlled study was conducted on children aged between 3-10 years diagnosed with ASD at PSRD hospital having Different severity levels. DTT was provided through a video training program using digital technology with informed consent from their caregivers/parents. The sample size was 10. Both groups contain 5 participants. The treatment group will be trained on DTT through the video training program. Sessions were conducted thrice a week for 45 minutes. The duration of the experiment was 12 weeks. The control group did not intervene with the video training program during the experiment. Pre & Post language assessment was done through British Picture Vocabulary Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 3-10 years.
* Clinically diagnosed children from Psychologists were taken for study who had 2-3 words in vocabulary or no vocabulary at all.
* Each group received 3 weekly sessions for 45 minutes for 12 weeks.
* Video training was given through animated videos.

Exclusion Criteria:

* Children with any comorbidities e.g. Intellectual Disability, Cerebral Palsy, Attention Deficit Hyperactive Disorder, Down's Syndrome and Hearing Impaired children will exclude from this study.
* Children diagnosed with severe autism.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
British Picture Vocabulary Scale | 3 months
  It helps you identify any delay in vocabulary development, even before children are in full-time education. BPVS3 is a one-to-one test in a simple and easy to administer format. For each question, you say a word and the pupil responds by selecting a picture from four options that best illustrates that word's meaning

CONTACTS AND LOCATIONS:
Overall Officials: Shahzadi Arshad, MS SLP, Principal Investigator — Pakistan Society for Rehabilitation of differently abled
Locations (1):
- Pakistan society for rehabilitation of differently abled, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No